CLINICAL TRIAL: NCT05013333
Title: Post-Approval Study for AED 3 With Uni-padz
Brief Title: AED 3 Post-Approval Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zoll Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 47701
Record Dates: First submitted 2021-08-16; First posted 2021-08-19 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Cardiac Arrest, Out-Of-Hospital
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- AED 3 with Uni-padz (Other)
  Interventions: Device: AED 3 with Uni-padz

INTERVENTIONS:
Device: AED 3 with Uni-padz — Use of AED 3 with Uni-padz by lay rescuer

SUMMARY:
Demonstrate appropriate CPR sensor placement on pediatric and adult patients and demonstrate delivery of appropriate energy level of shocks to pediatric and adult patients.

ELIGIBILITY:
Inclusion Criteria:

* Suspected out-of-hospital cardiac arrest
* Use of ZOLL AED 3 public-access defibrillator (running software v.1.03.602 or newer (US) or v. 6.03.006 or newer(OUS)) with Uni-padz III
* Unconsciousness
* Absence of breathing
* Absence of pulse and other signs of circulation

Exclusion Criteria:

* Pre-existing Do Not Attempt Resuscitation (DNAR) orders
* No evidence of cardiac arrest

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2021-03-30 (Actual); Primary Completion 2029-02-28 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
CPR sensor placement | Procedure (At time of device placement)
  Rate of appropriate placement of the CPR electrodes and compression sensor
Selection of adult or pediatric mode | Procedure (At time of device placement)
  Rate of appropriate selection of child mode by pressing "Child Mode" button or adult mode by not pressing "Child Mode" button determined by energy level of first shock

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University at Buffalo, Buffalo, New York
  - Colonie EMS, Latham, New York

IPD SHARING:
Plan to Share IPD: No